CLINICAL TRIAL: NCT04776603
Title: A Comparison of the Accuracy of Many Different Toric Intraocular Lens Formulas
Brief Title: A Comparison of the Accuracy of Toric Intraocular Lens Formulas
Status: Completed | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Other Study IDs: Toric-CPJ
Record Dates: First submitted 2020-11-30; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Astigmatism
Keywords: calculators; cataract; intraocular lens power; toric
MeSH Terms: conditions — Astigmatism; Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: group 1 includes patients who axial length(AL)<26mm
- Group 2: group 2 includes patients who axial length（AL）≥26mm

SUMMARY:
To compare the accuracy of the Abulafia-Koch, the Barrett, the Barrett Post ,the EVO , the new Holladay with total surgical-induced astigmatism, the Kane and and the Næser-Savini toric intraocular lens (IOL) power formulas using a large database of toric IOL refractive outcomes

DETAILED DESCRIPTION:
To compare the accuracy of the Abulafia-Koch, the Barrett, the Barrett Post ,the EVO , the new Holladay with total surgical-induced astigmatism, the Kane and and the Næser-Savini toric intraocular lens (IOL) power formulas using a large database of toric IOL refractive outcomes.Retrospective consecutive case series.One hundred seventy-two eyes of 172 patients who had a toric IOL inserted during surgery.One eligible eye from patients having uncomplicated cataract surgery with insertion of an Alcon SN6AT(2-9) IOL (Alcon Laboratories, Inc, Fort Worth, TX) from 1 surgeon were included in the study. pre-operative were measured using either the IOLMaster 500 or 700 (Carl Zeiss Meditec AG, Jena, Germany). Using vector calculation, the predicted postoperative refractive astigmatism was calculated for each formula. This was compared with the actual postoperative refractive astigmatism to give the prediction error.

ELIGIBILITY:
Inclusion Criteria:

* uncomplicated cataract surgery with a temporal clear corneal incision,with preoperative biometry using either the IOLMaster 500 (softwareversions 5.5 and 7.7) or 700 (software version 1.50; Carl Zeiss Meditec AG, Jena, Germany)
* subjective manifest refraction performed by any of the orthoptists in the practice and measurement of the actual postoperative axis of the IOL alignment performed in the same visit an average of 1 or 3months after surgery.

Exclusion Criteria:

* any corneal disease (keratoconus, other ectasia, pterygium, or previous trauma);
* previous ophthalmic operations, including laser vision correction, vitrectomy, pterygium surgery, penetrating glaucoma surgery, or scleral buckling procedures
* intraoperative or postoperative complications
* postoperative corrected distance visual acuity worse than 6/9

Ages: 21 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent cataract surgery at Eye hospital of Wenzhou Medical University,with insertion of the Alcon SN6AT(2-9) IOL(Alcon Laboratories, Inc, Fort Worth, TX)
Sampling Method: Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
A Comparison of the Accuracy of Toric Intraocular Lens Formulas | 5 years
  percentage of eyes with a prediction error within ±0.50 diopter (D)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang, China

REFERENCES:
- [Background] Abulafia A, Koch DD, Wang L, Hill WE, Assia EI, Franchina M, Barrett GD. New regression formula for toric intraocular lens calculations. J Cataract Refract Surg. 2016 May;42(5):663-71. doi: 10.1016/j.jcrs.2016.02.038. PMID 27255241
- [Result] Kane JX, Connell B. A Comparison of the Accuracy of 6 Modern Toric Intraocular Lens Formulas. Ophthalmology. 2020 Nov;127(11):1472-1486. doi: 10.1016/j.ophtha.2020.04.039. Epub 2020 May 1. PMID 32371252